CLINICAL TRIAL: NCT00463112
Title: Effect of Diet Plus Sibutramine on Hormonal and Metabolic Features in Overweight and Obese Women With PCOS: a Randomized, 24-Week Study
Brief Title: Effect of Diet Plus Sibutramine on Hormonal and Metabolic Features in Overweight and Obese Women With PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 511/8-1-04
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2003-12

CONDITIONS: Obesity; Polycystic Ovary Syndrome
Keywords: Obesity; Polycystic Ovary Syndrome; weight loss; Hyperadrogonemia; Sibutramine
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome; Weight Loss | interventions — sibutramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sibutramine

SUMMARY:
Studies on the effect of sibutramine, an anti-obesity drug, on hormonal and metabolic features of women with polycystic ovary syndrome (PCOS) are lacking.

The objective of this study is to examine the effect of sibutramine plus hypocaloric diet on body composition, hormonal and metabolic parameters and insulin resistance in obese patients with PCOS.

Overweight and obese women with PCOS were placed in a hypocaloric diet plus sibutramine (10 mg/day) for the first month and then on a hypocaloric diet plus sibutramine (10 mg/day) or hypocaloric diet only for the subsequent 6 months.

The main outcome measures are: Body composition, hormonal and metabolic features and insulin sensitivity (OGTT) at baseline, at 3 and 6 months of treatment.

DETAILED DESCRIPTION:
The Polycystic Ovary Syndrome (PCOS) is one of the most common hormonal disorders in women of reproductive age. As a syndrome it has multiple components, such as reproductive (chronic anovulation and infertility), metabolic and cardiovascular. Although lean women present PCOS, obesity is one of the main manifestations of the syndrome. Androgen excess and insulin resistance underline much of the clinical and metabolic features of the syndrome.

Recent evidence suggests that PCOS patients have a substantial risk for the development of metabolic and cardiovascular abnormalities similar to those presented in the metabolic syndrome. Obesity, particularly of the abdominal type, is presented in approximately half of the women with PCOS, although several studies have shown that percentage can vary from 30% to 75%. Several studies have demonstrated that obesity in women with PCOS enhances the clinical and metabolic abnormalities of the syndrome, since obese women with PCOS have more profound insulin resistance or type 2 DM,dyslipidemia and cardiovascular disease's risk, and greater level of androgens due to low SHBG levels.

A modest weight loss (<5% or even 5-10% of initial body weight) has been shown to improve ovulation frequency and conception, to reduce miscarriage, hyperlipidemia, hypertension, hyperglycemia and insulin resistance in women with PCOS. There are only a few studies on the effect of anti-obesity drug administration in obese and overweight women with PCOS. To the authors' best knowledge, the effect of sibutramine, a serotonin and noradrenaline reuptake inhibitor (SNRI) approved as antiobesity drug, has been studied in only one study with obese women with PCOS. Given this lack of information, the aim of the present study was to investigate any additional effect of sibutramine combined with a hypocaloric diet on body composition, hormonal and lipids parameters and insulin resistance in obese women with PCOS.

Study's design The study was prospective, open label, randomized, comparative trial. The study design included 3 periods; a screening period in order to confirm the diagnosis of PCOS, a lead-in period (4 weeks duration) that all patients were prescribed 10mg/day sibutramine plus a 600 kcal deficient diet, and a treatment period (for the subsequent 6 months) that subjects were randomized in a 2:1 ratio to the S group (10 mg/day of Sibutramine plus hypocaloric diet) and the D group (hypocaloric diet only). Diet was based on the individualized basal metabolic rate as defined by the Harris-Benedict's equation adjusted for moderate physical activity. Before entering the lead-in period all subjects were prescribed an energy-restricted diet containing 50% as carbohydrate, 30% as fat (10% saturated), and 20% as protein. After randomization, subjects were advised not to modify their eating habits throughout the study period.

The randomization was performed using sealed envelopes prepared in advance of the study by a research associate not involved in the study. A randomisation table was created using blocks of 3 numbers with all possible combinations. A random number generator has been used to create balance between the treatment groups.

Clinical measures Body weight, waist circumference and fasting blood samples for total testosterone (T), Sex Hormone Binding Globulin (SHBG), dehydroepiandrosterone sulfate (DHEAS), androstenedione (Δ4Α), 17a-hydroxyprogesterone, follicle stimulating hormone (FSH), luteinising hormone (LH), thyroid stimulating hormone (TSH), total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), glucose, and insulin were taken at baseline as well as at 3 and 6 months of treatment. At the same period, an Oral Glucose Tolerance Test (OGGT) with 75-g glucose was performed.

Blood samples were collected between 08:30 and 09:00 a.m., after an overnight fast, and during the follicular phase of women's menstrual cycle. Monthly, subjects' body weight was measured, adverse events, heart rate, blood pressure, and study drug compliance were determined and a pregnancy urine test was performed. Body weight was always determined at morning hours with subjects in light clothes.

ELIGIBILITY:
Inclusion Criteria:

* overweight and obese women with PCOS

Exclusion Criteria:

* Nonclassical 21-hydroxylase deficiency, hyperprolactinemia, adrenal or ovarian tumor and Cushing's disease, hypertension, thyroid dysfunction, overt diabetes mellitus and concomitant treatment such as antihypertensive drugs, SSRI or other SNRI drug, oral contraceptive pills or any other antiandrogen treatment (cyproterone acetate, spirolactone, LHRH agonist) and insulin sensitizing agents (metformin, pioglitazone, roziglitazone) that may interact with insulin sensitivity and lipid profile.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2004-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
weight loss

SECONDARY OUTCOMES:
FAI, insulin resistance and other metabolic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Dimos Florakis, MD, Principal Investigator — Divison of Endocrinology and Human Reproduction, Second Department of Obstetrics and Gynecology, Medical School, Aristotle University of Thessaloniki, Greece
Locations (1):
- Hippocratio General Hospital, Thessaloniki, Thessaloniki, Greece